CLINICAL TRIAL: NCT03959072
Title: Cardiac Cath Lab Staff Radiation Exposure During Chronic Total Occlusion PCI: CorPath GRX vs. Manual
Brief Title: Cardiac Cath Lab Staff Radiation Exposure
Acronym: SAFE-T
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision due to lower than anticipated enrollment
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 104-08553
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Robotic Chronic Total Occlusion PCI: The procedure will be randomized in a 1:1 fashion to either CorPath GRX robotic-assisted Chronic Total Occlusion PCI or conventional manual Chronic Total Occlusion PCI.
  Interventions: Device: Robotic CTO PCI
- Conventional (manual) Chronic Total Occlusion PCI: The procedure will be randomized in a 1:1 fashion to either CorPath GRX robotic-assisted Chronic Total Occlusion PCI or conventional manual Chronic Total Occlusion PCI.
  Interventions: Procedure: Conventional (Manual) CTO PCI

INTERVENTIONS:
Device: Robotic CTO PCI — Randomized to robotic CTO PCI.
  Other Names: CorPath GRX System
  Groups: Robotic Chronic Total Occlusion PCI
Procedure: Conventional (Manual) CTO PCI — Randomized to manual CTO PCI.
  Groups: Conventional (manual) Chronic Total Occlusion PCI

SUMMARY:
The objective of this randomized safety and observational study is to demonstrate CorPath GRX chronic total occlusion PCI is safe, and that Cardiac Catheterization Laboratory staff have no additional exposure to radiation when compared to conventional manual chronic total occlusion PCI procedures without added procedure time.

DETAILED DESCRIPTION:
This is prospective, dual-arm, randomized, multi-center, observational study comparing patient outcomes and staff radiation exposure in chronic total occlusion PCI procedures through 48 hours post procedure or hospital discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* CTO lesion, successfully crossed with conventional manual techniques;
* The Investigator deems the procedure appropriate for robotic-assisted CTO PCI with the CorPath GRX System;
* Individual monitoring of radiation dose, using the pocket dosimeter, was initiated at start of procedure;
* The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Failure/inability/unwillingness to provide informed consent, or
* Cardiogenic Shock; or
* Perforation which requires treatment (e.g. covered stent, coil and other embolization techniques, or pericardiocentesis).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects >18 years of age with symptoms suggestive of ischemic heart disease, with TIMI grade 0 flow and a lesion that is thought to be present for more than 3 months.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 48 hours
  Defined as successful CTO PCI revascularization with achievement of <30% residual diameter stenosis (visual estimate) within the treated segment and restoration of antegrade TIMI grade 3 flow, without in-hospital major adverse events (MAE).
In-hospital Major Adverse Events (MAE) | 48 hours
  Number of MAE events that occurs within 48 hours of the CTO PCI procedure or hospital discharge, whichever occurs first.

SECONDARY OUTCOMES:
Operator Radiation Exposure | Procedure
  Cumulative dose the physician receives as recorded from electronic pocket dosimeter during procedure.
Staff Radiation Exposure | Procedure
  Cumulative dose the staff receives as recorded from electronic pocket dosemeter during procedure.
Patient Radiation Exposure | Procedure
  DAP (dose-area-product) and cumulative dose/air kerma as recorded during the procedure
Fluoroscopy Time | Procedure
  Total fluoroscopy (min.) utilized during the procedure as recorded by an Imaging System.

CONTACTS AND LOCATIONS:
Overall Officials: William Lombardi (Acting), MD, Principal Investigator — University of Washington; William Nicholson (Emeritus), MD, Principal Investigator — WellSpan York Hospital
Locations (3):
- United States (3):
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - WellSpan York Hospital, York, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available 12 months after study completion.

REFERENCES:
- [Background] Hirshfeld JW Jr, Balter S, Brinker JA, Kern MJ, Klein LW, Lindsay BD, Tommaso CL, Tracy CM, Wagner LK, Creager MA, Elnicki M, Lorell BH, Rodgers GP, Weitz HH; American College of Cardiology Foundation; American Heart Association/; HRS; SCAI; American College of Physicians Task Force on Clinical Competence and Training. ACCF/AHA/HRS/SCAI clinical competence statement on physician knowledge to optimize patient safety and image quality in fluoroscopically guided invasive cardiovascular procedures: a report of the American College of Cardiology Foundation/American Heart Association/American College of Physicians Task Force on Clinical Competence and Training. Circulation. 2005 Feb 1;111(4):511-32. doi: 10.1161/01.CIR.0000157946.29224.5D. No abstract available. PMID 15687141
- [Background] Klein LW, Miller DL, Balter S, Laskey W, Haines D, Norbash A, Mauro MA, Goldstein JA; Joint Inter-Society Task Force on Occupational Hazards in the Interventional Laboratory. Occupational health hazards in the interventional laboratory: time for a safer environment. Catheter Cardiovasc Interv. 2009 Feb 15;73(3):432-8. doi: 10.1002/ccd.21801. PMID 19214981
- [Background] Miller DL, Schueler BA, Balter S; National Council on Radiation Protection and Measurements; International Commission on Radiological Protection. New recommendations for occupational radiation protection. J Am Coll Radiol. 2012 May;9(5):366-8. doi: 10.1016/j.jacr.2012.02.006. No abstract available. PMID 22554637
- [Background] Ciraj-Bjelac O, Rehani MM, Sim KH, Liew HB, Vano E, Kleiman NJ. Risk for radiation-induced cataract for staff in interventional cardiology: is there reason for concern? Catheter Cardiovasc Interv. 2010 Nov 15;76(6):826-34. doi: 10.1002/ccd.22670. PMID 20549683
- [Background] Vano E, Kleiman NJ, Duran A, Romano-Miller M, Rehani MM. Radiation-associated lens opacities in catheterization personnel: results of a survey and direct assessments. J Vasc Interv Radiol. 2013 Feb;24(2):197-204. doi: 10.1016/j.jvir.2012.10.016. Epub 2013 Jan 28. PMID 23369556
- [Background] Mahmud E, Naghi J, Ang L, Harrison J, Behnamfar O, Pourdjabbar A, Reeves R, Patel M. Demonstration of the Safety and Feasibility of Robotically Assisted Percutaneous Coronary Intervention in Complex Coronary Lesions: Results of the CORA-PCI Study (Complex Robotically Assisted Percutaneous Coronary Intervention). JACC Cardiovasc Interv. 2017 Jul 10;10(13):1320-1327. doi: 10.1016/j.jcin.2017.03.050. PMID 28683937

DOCUMENTS (1):
  • Study Protocol (2020-02-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03959072/Prot_001.pdf